CLINICAL TRIAL: NCT01248715
Title: Title: Effectiveness of Empiric Antiviral Treatment for Hospitalized Community Acquired Pneumonia During the Influenza Season (U18)
Brief Title: Rapid Empiric Treatment With Oseltamivir Study (RETOS)
Acronym: RETOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RETOS
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Influenza; Pneumonia
Keywords: pneumonia, bacterial; pneumonia, viral; respiratory tract infections; oseltamivir, therapeutic use
MeSH Terms: conditions — Influenza, Human; Pneumonia; Pneumonia, Bacterial; Pneumonia, Viral; Respiratory Tract Infections | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oseltamirvir (Experimental): These patients will receive early oseltamivir plus current, standard empiric antibacterial therapy.
  Interventions: Drug: oseltamivir
- Standard of care (No Intervention): These patients will be treated with the current, standard care, including currently recommended antibiotics or antiviral therapy based on national recommendations from the IDSA/ATS guidelines for management of hospitalized patients with CAP and ACIP antiviral use guidelines for hospitalized patients with confirmed of suspect influenza, per clinician discretion. In addition these patients with have a NP swab collected for influenza PCR testing and clinical information will be extracted from the medical record.

INTERVENTIONS:
Drug: oseltamivir — These patients will receive early (within 8-12 hours of admission, no later than 24 hours after admission) oseltamivir plus current, standard empiric antibacterial therapy based on national recommendations from the IDSA/ATS guidelines for management of hospitalized patients with CAP (2). Anti-influenza therapy will be given using oseltamivir at a dose of 75 mg twice daily. The oseltamivir dose will be adjusted in patients with renal insufficiency according to the package insert. Duration of antiviral therapy will be for a minimum of 5 days for patients with evidence of early clinical improvement and prolonged depending on clinical stability
  Other Names: Tamiflu
  Arms: Oseltamirvir

SUMMARY:
Current guidelines recommend early initiation of empiric antibiotic therapy to cover typical and atypical bacteria that may cause community-acquired pneumonia (CAP). Influenza antiviral therapy in patients with suspected or confirmed influenza. However, many clinicians do not suspect influenza among patients with CAP or other acute lower respiratory tract illness (LRTI) and often do not test for influenza. Additionally, results from currently available diagnostic tests for influenza may be delayed and several tests have low sensitivity and will give false negative results. Thus, anti-influenza treatment for patients with hospitalized influenza CAP and LRTI is frequently initiated late if at all. There is an association between delayed time to administration of empiric antibiotic therapy with increased clinical failure and mortality. As a result, empiric antibiotic therapy for patients with suspect CAP is begun within 4 - 6 hours of hospitalization. This has recently been demonstrated for delayed antiviral treatment as well. We hypothesize that, as happens with early empiric antibiotics for bacterial CAP, a standardized approach of adding early empiric anti-influenza therapy during the influenza season to hospitalized patients with suspect CAP and LRTI will improve clinical outcomes of patients with influenza associated CAP and LRTI.

To test our hypothesis we plan a prospective, randomized, multicenter clinical trial of hospitalized patients with acute LRTI, including suspect CAP, during . If early anti-influenza medications were not included on the patients admission orders, patients will be randomized to standard care, including empiric antibacterial therapy as recommended by ATS/IDSA guidelines plus standard influenza diagnostics and treatment (Standard of care) versus early initiation of empiric antiinfluenza therapy plus standard care, e.g. empiric antibacterial (oseltamivir group). The primary study outcome will be development of clinical failure and selected clinical outcomes during the 30 days after enrollment. Other clinical outcomes that will be compared between study groups include time to clinical stability, duration of hospitalization, development of cardiovascular events, re-hospitalization, short-term mortality (30 days), and long-term mortality (1 year). The secondary study outcome will be the cost-effectiveness of the intervention.

DETAILED DESCRIPTION:
This will be both a prospective, randomized, unblinded clinical study of hospitalized patients with acute LRTI admitted in one of four institutions in Louisville, KY (rapid empiric treatment with oseltamivir study[RETOS]) and a prospective observation study to describe influenza LRTI (Flu LRTI study). All hospitalized patients with acute LRTI will be invited to participate in one of the arms of study. If the admitting clinician does not order oseltamivir or zanamivir at the time of hospital admission, the patient is eligible for randomization into Group A (standard clinical care, including empiric antibiotics and anti-influenza drugs at the clinician discretion) or Group B (oseltamivir administered to the patient within 24 hours of admission, ideally within 8-12 hours of admission, plus empiric antibiotics).

Patients will be enrolled from one of four hospitals, the University of Louisville Hospital, Veterans Affairs Medical Center of Louisville, Norton Hospital of Louisville, and Jewish Hospital of Louisville. Eligible patients will be identified primarily in the Emergency Departments of all four hospitals and evaluated for inclusion/exclusion criteria after hospital admission orders are written. Patients will be enrolled only during the influenza season. For this study, the influenza season is defined as December 1st until May 1st, unless surveillance data suggests that influenza viruses are circulating earlier or have stopped circulating.

For all three study groups, diagnosis of influenza will be based on nucleic acid amplification through polymerase chain reaction (PCR). At the time of enrollment into the study, a nasopharyngeal swab will be obtained for PCR. The University of Louisville Infectious Diseases Reference Laboratory has extensive experience using molecular techniques for the diagnosis of respiratory pathogens and will test batched specimens at monthly intervals. In addition, we will collect the results from tests done for routine care and bacterial or virus isolates identified during routine care for further characterization.

The management of patients in Group A and Group B will be different only in regard to early empiric anti-influenza therapy. All other aspects of the management of these patients will be in compliance with national guideline recommendations from IDSA/ATS (2). Patients in Group A may have antiviral therapy started later in hospitalization or not treated at all. The study will not interfere with Group A patient care.

A 1:1 randomization ratio within the two study arms is planned for EOS. A pre-defined randomization chart will be designed in order to have the randomization process Internet-based. The randomization table will be accessible by the project manager as a back up in the event that any problem occurs with the Internet or the computerized system.

We will attempt to begin oseltamivir within 8 - 12 hours after hospital admission, and no later than 24 hours. The study nurse will facilitate receipt of early oseltamivir treatment for the consented patient in collaboration with the hospital pharmacies. The time of oseltamivir administration will be recorded for all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

For oseltamivir and standard of care groups:

* 18 years of age or older
* No oseltamivir or zanamivir ordered in hospital admission orders
* Meets criteria for acute LRTI
* Signed informed consent.

Exclusion Criteria:

For oseltamivir and standard of care groups:

* Oseltamivir or zanamivir ordered in hospital admission orders
* Patients hospitalized for the LRTI for more than 24 hours before enrollment into the trial.
* Patients with mental conditions who are unlikely to comply with the study protocol and who cannot give informed consent and have no guardian or proxy.
* Patients who have had severe allergic reactions such as anaphylaxis or serious skin reactions such as toxic epidermal necrolysis, Stevens-Johnson syndrome, or erythema multiforme to any component of oseltamivir (TAMIFLU).
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1107 (Actual)
Dates: Start 2010-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Ramirez, MD, Principal Investigator — University of Louisville
Locations (5):
- United States (5):
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Rex Robley VA Medical Center, Louisville, Kentucky
  - Baptist Hospital East, Louisville, Kentucky

REFERENCES:
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Derived] Wiemken TL, Furmanek SP, Carrico RM, Peyrani P, Hoft D, Fry AM, Ramirez JA. Effectiveness of oseltamivir treatment on clinical failure in hospitalized patients with lower respiratory tract infection. BMC Infect Dis. 2021 Oct 27;21(1):1106. doi: 10.1186/s12879-021-06812-2. PMID 34702188
- [Derived] Wiemken TL, Jala VR, Kelley RR, Peyrani P, Mattingly WA, Arnold FW, Cabral PW, Cavallazzi R, Haribabu B, Ramirez JA. The upper respiratory tract microbiome of hospitalised patients with community-acquired pneumonia of unknown aetiology: a pilot study. Pneumonia (Nathan). 2015 Dec 1;6:83-89. doi: 10.15172/pneu.2015.6/682. eCollection 2015. PMID 31641582
- [Derived] Ramirez J, Peyrani P, Wiemken T, Chaves SS, Fry AM. A Randomized Study Evaluating the Effectiveness of Oseltamivir Initiated at the Time of Hospital Admission in Adults Hospitalized With Influenza-Associated Lower Respiratory Tract Infections. Clin Infect Dis. 2018 Aug 16;67(5):736-742. doi: 10.1093/cid/ciy163. PMID 29659754
- See also: National Center for Health Statistics — http://www.cdc.gov/nchs/data/hus/hus06.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oseltamirvir | Standard of Care
Started | 556 | 551
Completed | 55 | 41
Not Completed | 501 | 510
Not completed — Not influenza positive | 501 | 510

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oseltamirvir | Standard of Care | Total
Number analyzed (Participants) | 55 | 41 | 96
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [41.5 to 84.5] | 60 [43 to 77] | 61.7 [42.1 to 81.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 32 | 18 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 41 | 96
Nursing home Resident [Count of Participants; unit: Participants] | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Failure (Failure to Reach Clinical Stability)
Description: Number of subject that showed lack of clinical improvement within 7 days. Criteria for clinical improvement include no fever; white blood cell count decreases, or increases in the case of leukopenia, to more than 10% from the prior day; the evaluation of signs and symptoms of CAP to define when the patient is subjectively better, and the patient is able to tolerate food by mouth.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
Participants | 6 | 2
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .460, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Participants to Transfer to ICU After 24 h
Description: Number of subjects that were transfered to an intensive care unit (ICU) after 24 hours of hospitalization. A patient transferred to ICU within 24 hours of admission was considered as a direct admission to ICU and not meeting criteria for clinical failure.
Time Frame: 24 h
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
Participants | 2 | 2
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .9999, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Participants That Required Re-hospitalization
Description: Participants that were re-hospitalized within 30 days after enrollment.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
Participants | 5 | 5
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .732, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Number of Participants That Had Short-term Mortality
Description: Number of subjects who died within 30 days of enrollment
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
Participants | 2 | 1
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .9999, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Days to Reach Clinical Stability
Description: Time to clinical improvement. The criteria for clinical improvement were followed during the first week from the day of admission and defined as follows: a) improvement of signs and symptoms of LRTI reported by patient b) afebrile for at least 8 hours, c) decrease in white blood cell count to more than 10% from the prior day, and d) able to tolerate oral feeding. A patient was considered clinically improved on the day that these four criteria were all met.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
days | 2 [0 to 4] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .685, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Length of Hospital Stay
Description: Duration of hospitalization calculated as the day of discharge minus the day of admission.
Time Frame: through study completion, up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
days | 4 [0 to 8] | 4.5 [1.5 to 7.5]
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .796, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Participants With Hospital Mortality.
Description: Number of subjects who died while hospitalized
Time Frame: through study completion, up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamirvir | Standard of Care
Number analyzed (Participants) | 55 | 41
Participants | 1 | 1
Statistical Analysis 1: Comparison: Oseltamirvir vs Standard of Care; Test type: Superiority; p = .9999, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Oseltamirvir | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/55 | 1/41
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/41
Other Adverse Events (participants affected / at risk) | 0/55 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamirvir (N=55) | Standard of Care (N=41)
Cardiovascular event (Cardiac disorders) | 0 (0) | 1 (1) — Subject was readmitted to the hospital with chest pain and congestive heart failure not related to the drug.

LIMITATIONS AND CAVEATS:
The primary limitation of our study that we were not able to reach the number of patients that were estimated in the sample size calculation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes